CLINICAL TRIAL: NCT03827317
Title: HERPET: A Mechanistic Non-Invasive Imaging Study of HER2 Expression in Breast Cancer Using [18F]GE-226 Positron Emission Tomography
Brief Title: HERPET- A Novel PET Imaging Study of HER2 in Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government); University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015-004027-31
Record Dates: First submitted 2019-01-17; First posted 2019-02-01 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
Keywords: HER2; imaging; PET; positron emission tomography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Non-randomised cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HER2 positive metastatic breast cancer (Other): 8 HER2 positive patients (determined using the most recent biopsy) will be recruited. Dynamic [18F]GE-226 PET imaging over 90 minutes, radial artery sampling will be performed to establish the pharmacokinetic profile of [18F]GE-226 and hence determine the optimal imaging time point for [18F]GE-226 PET scans. Tumour uptake in individual metastases (and the target lesion) will be reported. Uptake will be compared between HER2 positive and negative tumours.
  Interventions: Radiation: [18F]GE-226
- HER2 negative metastatic breast cancer (Other): 8 HER2 negative patients (determined using the most recent biopsy) will be recruited. Dynamic [18F]GE-226 PET imaging over 90 minutes, radial artery sampling will be performed to establish the pharmacokinetic profile of [18F]GE-226 and hence determine the optimal imaging time point for [18F]GE-226 PET scans. Tumour uptake in individual metastases (and the target lesion) will be reported. Uptake will be compared between HER2 positive and negative tumours.
  Interventions: Radiation: [18F]GE-226

INTERVENTIONS:
Radiation: [18F]GE-226 — [18F]GE-226 is a radiolabelled Affibody® tracer which binds to the HER2 receptor with high affinity at a different epitope than trastuzumab. The active molecule is a 61 amino acid peptide that is modified site-specifically with one fluorobenzaldehyde molecule at the C-terminal.

SUMMARY:
This mechanistic study will be the first study to assess the efficacy of [18F]GE-226 to target HER2 expression in patients with metastatic breast cancer. The study will establish the pharmacokinetics of [18F]GE-226 and the optimum time-point for performing static scans in this patient population.

DETAILED DESCRIPTION:
Objectives

Primary:

* To determine the uptake in tumour lesions and normal tissue of [18F]GE-226 and compare the difference between patients with HER2 positive and HER2 negative lesions. Uptake will be quantified by semi-quantitative (SUV, AUC) and fully quantitative parameters (Ki in the case of irreversible uptake, and binding potential in the case of reversible uptake)
* To determine the optimal imaging time point for [18F]GE-226

Secondary:

* To determine the safety and toxicity of [18F]GE-226 PET in humans
* To determine if [18F]GE-226 can distinguish between HER2 amplified and HER2 non-amplified breast tumours
* To determine the metabolism of [18F]GE-226 in human subjects

Exploratory:

• To explore circulating biomarkers that may be related to [18F]GE-226 uptake and to investigate if treatment modulates [18F]GE-226

Endpoints

Secondary:

* Safety and toxicity of [18F]GE-226 measured by adverse events from administration of [18F]GE-226 injection throughout the study period, and clinically significant changes from baseline measurements in serum biochemistry, haematology, coagulation, immunology, urinalysis, vital signs, ECG, injection site and physical examination findings.
* The association between [18F]GE-226 tumour uptake and standard HER2 pathological testing (HER2 amplified and HER2 non-amplified breast tumours)
* Proportion of metabolised [18F]GE-226 at scheduled time-points compared to baseline
* Normal tissue uptake of [18F]GE-226 will be quantified in the appropriate regions depending on the field of view.

Exploratory:

• To perform preliminary biodistribution analysis, to compare [18F]GE- 226 uptake to [18F]FDG uptake in tumour lesion

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with a histological diagnosis of breast cancer with known HER2 status ((8 positive and 8 negative).
2. Written informed consent prior to admission in the study.
3. Target lesion diameter of ≥15mm that has not been previously irradiated.
4. Female patients aged ≥ 18 years of age.
5. For all patients: histologically confirmed locally advanced/metastatic breast cancer with a biopsy within the last 12 months confirming HER2 status by either immunohistochemistry (IHC), Silver In Situ Hybridization (SISH) or Fluorescent In Situ Hybridization (FISH).
6. ECOG performance status 0-2
7. Negative urine pregnancy test (within 2 hours prior to injection of imaging agent) in women of child bearing age and willingness to use contraception (barrier, abstinence, non-hormonal) for 3 weeks after injection of [18F]GE-226
8. Life expectancy > 3 months
9. Adequate organ function as defined by

   * Hb≥10g/L
   * WBC≥3.0 x 109/L
   * PLT≥80 x 109/L
   * Serum creatinine ≤1.4mg/dl
   * SGOT and SGPT ≤2 x ULN
   * Total bilirubin ≤ 2 x ULN or 3.0 mg/dl in patients with Gilbert's syndrome
10. Patients must have been appropriately staged using FDG-PET within 42 days of study entry and additional imaging according to local standard of care

Exclusion Criteria:

1. Pregnant or lactating women.
2. History of cardiac disease (myocardial infarction, arrhythmias requiring therapy, symptomatic valvular disease, cardiomyopathy, or pericarditis).
3. Evidence of significant medical condition or laboratory finding which, in the opinion of the Investigator, makes it undesirable for the patient to participate in the trial.
4. Participants with severe claustrophobia or who are unable to lie flat or fit into the scanner (≥350 lbs (160 Kg)).
5. Prior use within 14 days of enrolment or concurrent therapy with any other investigational agent.
6. Patients classified as radiation workers
7. Patients on therapeutic doses of anticoagulants, or with a raised prothrombin time

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with a histological diagnosis of breast cancer with known HER2 status ((8 positive and 8 negative).
Enrollment: 24 (Estimated)
Dates: Start 2019-03-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumoral uptake of [18F]GE-226 in patients with breast cancer measured using semi-quantitative parameters | 24 months
  Tumoral uptake of [18F]GE-226 in patients with HER2 positive and HER2 negative breast cancer measured using SUV and AUC.
Tumoral uptake of [18F]GE-226 in patients with breast cancer measured using fully quantitative parameters | 24 months
  Tumoral uptake of [18F]GE-226 in patients with HER2 positive and HER2 negative breast cancer measured using Ki in the case or irreversible uptake, and binding potential in the case of reversible uptake.

SECONDARY OUTCOMES:
Adverse events of [18F]GE-226 injection | 0 hour, 48 hours
  Safety of [18F]GE-226 measured by adverse events from administration of [18F]GE-226 injection throughout the study period.
Serum biochemistry change from baseline measurement | 0 hour, 48 hours
  Safety of [18F]GE-226 injection measured by clinically significant changes from baseline measurements in serum biochemistry finding.
Haematology change from baseline measurement | 0 hour, 48 hours
  Safety of [18F]GE-226 injection measured by haematology change from baseline measurements.
Immunology change from baseline measurement | 0 hour, 48 hours
  Safety of [18F]GE-226 injection measured by clinically significant changes from baseline measurements in immunology
Urine change from baseline measurement | 0 hour, 48 hours
  Safety of [18F]GE-226 injection measured by clinically significant changes from baseline measurements in urine
EEG change from baseline measurement | 0 hour, 48 hours
  Safety of [18F]GE-226 injection measured by clinically significant changes from baseline measurements in ECG

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Kenny, MD FRCP PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No